CLINICAL TRIAL: NCT00547989
Title: Paravertebral Block, an Adjunct to General Anaesthesia for Breast Surgery?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC 05-105.5
Record Dates: First submitted 2007-10-18; First posted 2007-10-23 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Breast Cancer
Keywords: ASA class I and II
MeSH Terms: conditions — Breast Neoplasms | interventions — Bupivacaine; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): control
  Interventions: Drug: standard anaesthesia (bupivacaine)
- 2 (Experimental): PVB with ropivacaine and postoperative pump 5ml/h
  Interventions: Drug: additional pvb (ropivacaine) and elastomeric disposable infusion pump
- Experimental 1 (Experimental): PVB with ropivacaine, 10 patients included but not analysed
  Interventions: Drug: additional pvb (ropivacaine)

INTERVENTIONS:
Drug: standard anaesthesia (bupivacaine) — Local infiltration with bupivacaine and Piritramide and Paracetamol as postoperative analgesic, and ondansetron as required
  Arms: 1
Drug: additional pvb (ropivacaine) and elastomeric disposable infusion pump — Patients in group 2 will receive PVB with ropivacaine and postoperative pump 5ml/h.
  Arms: 2
Drug: additional pvb (ropivacaine) — Patients in group 1 will receive PVB with ropivacaine
  Arms: Experimental 1

SUMMARY:
Aim is to study if a paravertebral block as an adjunct to general anesthesia is a suitable technique for extended, one sided, breast surgery.

DETAILED DESCRIPTION:
Usually breast tumour surgery in the Academic Hospital Maastricht is performed under general anaesthesia. Perioperative pain management consists of paracetamol and naproxen preoperatively, opioids during surgery and local wound infiltration at the end of surgery with 10cc Bupivacaine 0.25%. Postoperative pain management consists of paracetamol, occasionally combined with Naproxen, and if necessary Piritramide 0.2 mg/kg i.m.

Alternatively there is the possibility to perform breast surgery under a thoracic paravertebral block (PVB) with or without general anesthesia.

A PVB according to Eason and Wyatt (1) can be performed preoperatively with insertion of an end-hole catheter T3-T4. With this technique we expect a better pain relief postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Extended mamma surgery one-sided
* ASA class I and II

Exclusion Criteria:

* All contra indications for local anaesthesia
* Coagulation disorders
* Infection
* Allergic reactions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2006-10; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
reduction of unplanned admissions and reduction of VAS score. | one week

SECONDARY OUTCOMES:
to determine the safety and performance (efficacy) of the technique and the investigational product. | one week

CONTACTS AND LOCATIONS:
Overall Officials: Esther Bouman, MD, Principal Investigator — azM
Locations (1):
- University Hospital, Maastricht, Netherlands